CLINICAL TRIAL: NCT05904184
Title: Comparison of the Clinical Effectiveness of Calcium Silicate-based Sealer and Epoxy Resin-based Sealer in Single-visit Root Canal Treatment
Brief Title: Comparison of Calcium Silicate-based Sealer and Epoxy Resin-based Sealer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Tran Ngoc Minh Duyen, University Post Graduated Student, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 452/HD-DHYD
Record Dates: First submitted 2023-02-23; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-02

CONDITIONS: Pulpitis - Irreversible; Pain, Postoperative
Keywords: Calcium silicate-based sealer; Epoxy resin-based sealer
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epoxy resin-based sealers (ERS) (Active Comparator): After root canal preparation, canal obturation was performed with Epoxy resin-based sealers (ERS)
  Interventions: Drug: Calcium silicate-based sealers (CSS)
- calcium silicate-based sealers (CSS) (Active Comparator): After root canal preparation, canal obturation was performed with Calcium silicate-based sealers (CSS)
  Interventions: Drug: Epoxy resin-based sealers (ERS)

INTERVENTIONS:
Drug: Epoxy resin-based sealers (ERS) — All teeth received one-visit endodontic treatment according to the treatment protocol of the Vietnamese Ministry of Health with the support of three-dimensional imaging equipment and an endodontic machine. After root canal preparation, obturation was performed using Epoxy resin-based sealers.
  Other Names: Epoxy resin-based cement
  Arms: calcium silicate-based sealers (CSS)
Drug: Calcium silicate-based sealers (CSS) — All teeth received one-visit endodontic treatment according to the treatment protocol of the Vietnamese Ministry of Health with the support of three-dimensional imaging equipment and an endodontic machine. After root canal preparation, obturation was performed using Calcium silicate-based sealers.
  Other Names: Calcium silicate-based cement
  Arms: Epoxy resin-based sealers (ERS)

SUMMARY:
Background: Sealers have been concerned with obturation. However, studies for assessing the effectiveness of endodontic treatment of sealer based on Calcium Silicate have been not much.

Objective: This study aimed to assess the effectiveness of endodontic treatment of sealer based on Calcium Silicate Methods: A prospective, single-blind, clinical trial was conducted from June 2020 to December 2020 with 42 irreversible pulpitis teeth by one clinician. The postoperative pain was assessed after root canal treatment using sealer based on Calcium Silicate and sealer based on Epoxy resin after 6 hours, 12 hours, 24 hours, 48 hours, 72 hours and 7 days and inconvenient symptoms were assessed after 7 days, 3 months and 6 months. t-test, Mann-Whitney and Wilcoxon analysis were applied.

Key words: obturation, sealer based on Calcium Silicate and sealer based on Epoxy resin

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* teeth diagnosed with irreversible pulpitis by electrical and thermal tests (+)
* had clinical symptoms like continuous or spontaneous pain, teeth exposed to sudden temperature changes, especially cold stimuli, causing sharp pain and persisting after stimulus removal
* these teeth must have healthy periodontal tissue and sufficient clinical teeth crown for isolation with a rubber dam

Exclusion criteria:

Patients with:

* Pregnant
* Have a systemic disease requiring antibiotics or have an allergic reaction
* Have maxillofacial pathology, cellulitis, occlusal trauma, and temporomandibular disorders, have endodontic periodontal lesions, periodontal abscesses
* Have taken a previous pain reliever within 24 hours

Tooth:

* Roots internally or externally resorbed, cracked or broken
* Have had failed endodontic treatment, or the root canal cannot be controlled for leakage
* No opposing teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity over time | after 6 hours, 12 hours, 24 hours, 48 hours, 72 hours and 7 days after treatment
  The investigator instructed patients on how to use the 170-mm Heft-Parker self-assessment scale to evaluate their pain intensity. Swelling, fistula, and sensitivity under biting pressure were classified as binary variables.
Change in pain relief over time | after 6 hours, 12 hours, 24 hours, 48 hours, 72 hours and 7 days after treatment
  The investigator instructed patients on how to use the 170-mm Heft-Parker self-assessment scale to evaluate their pain intensity. Swelling, fistula, and sensitivity under biting pressure were classified as binary variables.
Change in treatment outcome evaluation over time | 1 week, 3 months and 6 months after treatment
  Based on Strindberg's criteria of clinical symptoms, the treatment outcome evaluation was then expressed as success, failure, or uncertain depending on the presence of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sathorn C, Parashos P, Messer H. The prevalence of postoperative pain and flare-up in single- and multiple-visit endodontic treatment: a systematic review. Int Endod J. 2008 Feb;41(2):91-9. doi: 10.1111/j.1365-2591.2007.01316.x. Epub 2007 Oct 23. PMID 17956561
- [Background] El Mubarak AH, Abu-bakr NH, Ibrahim YE. Postoperative pain in multiple-visit and single-visit root canal treatment. J Endod. 2010 Jan;36(1):36-9. doi: 10.1016/j.joen.2009.09.003. PMID 20003932